CLINICAL TRIAL: NCT01290640
Title: In Vivo Comparison of Kinematics for Subjects Implanted With a Press Fit Condylar Sigma Rotating Platform or Fixed Bearing Total Condylar III Prothesis
Brief Title: Comparison of Kinematics for Subjects Implanted With a PFC Sigma Rotating Platform or Fixed Bearing TC3 Prosthesis
Acronym: PFC & TC3
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: Komistek AG 08-19-20; R011373360 (Other: UT Grant)
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Knee Prosthesis; Knee Arthroplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TC3 TKA: Subjects implanted with a DePuy fixed-bearing Total Condylar III (TC3) TKA
  Interventions: Device: DePuy fixed-bearing Total Condylar III (TC3) TKA
- PFC RP TC3 TKA: Subjects implanted with a DePuy PFC Rotating Platform TC3 TKA
  Interventions: Device: DePuy PFC Rotating Platform TC3 TKA

INTERVENTIONS:
Device: DePuy fixed-bearing Total Condylar III (TC3) TKA
  Groups: TC3 TKA
Device: DePuy PFC Rotating Platform TC3 TKA
  Groups: PFC RP TC3 TKA

SUMMARY:
The objectives of this study are four-fold:

1. To determine the three-dimensional, in vivo kinematics for subjects having either a fixed- or mobile-bearing Press Fit Condylar (PFC) Sigma Total Condylar III Prosthesis, comparing the in vivo kinematics to determine if one implant type leads to a benefit for the patient.
2. To determine if bearing mobility occurs in PFC Sigma Rotating Platform Total Condylar III Prosthesis under in vivo, weight-bearing conditions during multiple activities (gait, stair descent, deep knee bend and chair rise).
3. To determine if there is a correlation between in vivo kinematic data obtained using fluoroscopy, electromyography (EMG) and ground reaction force (GRF) data and determine if variability occurs between these two TKA types.
4. To determine if a clinical benefit is either visibly detected (video camera) or quantifiably determined (questionnaire) for either TKA type.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least three months post-operative.
2. Potential subjects will have a body weight of less than 250 lbs.
3. Candidates must have had a HSS score >90 post-operatively.
4. Patients must have passive flexion of at least 100.
5. All potential subjects will have a Press Fit Condylar (PFC) Rotating Platform Total Condylar III Prosthesis (Depuy Orthopaedics, Warsaw, IN) or fixed-bearing Total Condylar III Prosthesis.
6. Must be willing to sign both Informed Consent and HIPAA forms.

Exclusion Criteria:

1. Pregnant females.
2. Patients that do not meet study requirements.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects requiring total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Komistek, Ph D, Principal Investigator — The University of Tennessee; Douglas Dennis, MD, Principal Investigator — Colorado Joint Replacement, Porter Adventist Hosp
Locations (3):
- United States (3):
  - Porter Adventist Hospital, Denver, Colorado
  - Perkins Hall, Knoxville, Tennessee
  - Science and Engineering Research Facility, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 09/2011-12/2012, hospital
Groups:
- Subjects Implanted With a DePuy Fixed-bearing Total Condylar I: Subjects implanted with a DePuy fixed-bearing Total Condylar III (TC3) TKA
Period: Overall Study
Arm/Group | Subjects Implanted With a DePuy Fixed-bearing Total Condylar I | Subjects Implanted With a DePuy PFC Rotating Platform TC3 TKA
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PFC RP TC3 TKA | Subjects Implanted With a DePuy Fixed-bearing Total Condylar I | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (9.8) | 74.06 (10.1) | 72.5 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: In Vivo Linear Kinematics for Fixed-bearing and Rotating Platform (RP) TKA System During 4 Weight-bearing Activities.
Description: The values that were reported indicate the motion of the contact point from the start of the activity to the end of the activity. If the point translated forward (anteriorly) atop the tibial tray, the number was reported as positive. If the point traveled backwards (posteriorly) atop the tibial tray, the number was reported as negative.
Time Frame: March 2013
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Subjects With DePuy PFC Rotating Platform TC3 TKA | Subjects With DePuy PFC Fixed Bearing TC3 TKA
Number analyzed (Participants) | 10 | 12
Number analyzed (Implants) | 10 | 12
mm
  Lateral Anterior Posterior Deep Knee Bend | -3.51 (4.73) | -2.52 (1.92)
  Medial Anterior Posterior Deep Knee Bend | -1.68 (2.15) | -1.40 (1.43)
  Lateral Anterior Posterior Chair Rise | -10.31 (3.23) | 2.89 (3.64)
  Medial Anterior Posterior Chair Rise | -0.76 (3.95) | 1.02 (2.95)
  Lateral Anterior Posterior Gait | -0.88 (2.02) | -1.3 (1.8)
  Medial Anterior Posterior Gait | .70 (2.51) | -1.2 (1.5)
  Lateral Anterior Posterior Stair Descent | -8.18 (2.08) | -1.92 (2.46)
  Medial Anterior Posterior Stair Descent | -1.96 (3.22) | -1.71 (1.80)

2. Primary Outcome: In Vivo Angular Kinematics for Fixed-bearing and Rotating Platform (RP) TKA System During 4 Weight-bearing Activities.
Description: Angular kinematics for fixed bearing and rotating platform TKA system - Axial Rotation
  The values that were reported indicate the rotation of the femur atop the tibial tray from the start of the activity to the end of the activity. If the femur rotated externally (posterior rollback of the lateral condyle, generally pivoted about the medial condyle), the number was reported as positive. If the femur rotated internally (anterior slide of the lateral condyle, generally pivoted about the medial condyle), the number was reported as negative.
Time Frame: March 2013
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Implants
Arm/Group | Subjects With DePuy PFC Rotating Platform TC3 TKA | Subjects With DePuy PFC Fixed Bearing TC3 TKA
Number analyzed (Participants) | 10 | 12
Number analyzed (Implants) | 10 | 12
degrees
  Axial Rotation Deep Knee Bend | 8.35 (8.94) | 1.99 (4.00)
  Axial Rotation Chair Rise | 12.22 (8.29) | -2.42 (5.03)
  Axial Rotation Gait | 6.66 (6.37) | .13 (2.18)
  Axial Rotation Stair Descent | 8.16 (5.56) | .24 (4.17)

ADVERSE EVENTS:
Description: There were no adverse events encountered for any subjects in either group.
Arm/Group | Subjects Implanted With a DePuy PFC Rotating Platform TC3 TKA | Subjects Implanted With a DePuy Fixed-bearing Total Condylar I
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12

LIMITATIONS AND CAVEATS:
No limitations were encountered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No